CLINICAL TRIAL: NCT00830622
Title: A Targeted Cell Phone Intervention to Improve Patient Access to Care and Drug Adherence in Patients Taking Antiretroviral (ARV) Medications in Kenya
Brief Title: Cell Phone Intervention to Support Antiretroviral Therapy (ART) Adherence in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Nairobi (Other)
Responsible Party: Richard T. Lester, MD, FRCPC / Principal Investigator, Dept. of Medical Microbiology and Infectious Diseases, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H2007:037; CDC PEPFAR PHE KE.07.0045
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-01

CONDITIONS: HIV; AIDS; HIV Infections
Keywords: HIV/AIDS; Adherence; Antiretroviral Therapy, ART, ARV; Mobile phone, cell phone, telephone; Text message, SMS; Telemedicine; Africa; Resource-limited setting; Counseling, support; treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cell Phone Intervention: participant receives weekly SMS text message from the health care worker.
  Interventions: Other: Cell Phone Intervention
- 2 (No Intervention): SOC: Participant receives standard of care support but not weekly SMS text messages from the health care worker.

INTERVENTIONS:
Other: Cell Phone Intervention — Participant receives weekly SMS text messages from the health care provider.
  Arms: 1

SUMMARY:
A clinical study to evaluate the use of cell phones to support drug adherence and follow-up of patients taking antiretroviral therapy (ART) for treatment of HIV. The intervention involves health-care providers sending regular short-message-service (SMS) text messages to patients and following up their responses. The hypothesis is that the cell phone intervention will improve ART adherence and health outcomes compared with the current standard of care.

DETAILED DESCRIPTION:
This RCT study focuses on enrolling and following patients initiating ART. Note, a second parallel prospective cohort study enrolls and follows ART experienced patients who have already been taking ART for at least one year before and after the same intervention.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected and starting antiretroviral therapy
* Adequate (daily) access to a cell phone
* Intending to attend the enrollment clinic for 2 years
* Consent to participate

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Adherence to ART and HIV RNA suppression | 6,12 months
  Although many patients are seen every 3 months, study visits with questionnaires and viral load are completed at 0, 6, and 12 month scheduled follow-up visits.

SECONDARY OUTCOMES:
Retention | 6, 12 months
Quality of Life (SF-12) | 3, 6, 9, 12 months
Health (CD4, weight, progression to AIDS, all cause mortality) | 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lester, MD, FRCPC, Principal Investigator — University of Manitoba; Joshua Kimani, MBChB, Study Chair — University of Manitoba / University of Nairobi; Francis A Plummer, MD, FRCPC, Study Director — University of Manitoba
Locations (1):
- University of Nairobi Clinics, Nairobi, Kenya

REFERENCES:
- [Background] Lester R, Karanja S. Mobile phones: exceptional tools for HIV/AIDS, health, and crisis management. Lancet Infect Dis. 2008 Dec;8(12):738-9. doi: 10.1016/S1473-3099(08)70265-2. No abstract available. PMID 19022188
- [Background] Lester RT, Gelmon L, Plummer FA. Cell phones: tightening the communication gap in resource-limited antiretroviral programmes? AIDS. 2006 Nov 14;20(17):2242-4. doi: 10.1097/QAD.0b013e3280108508. No abstract available. PMID 17086071
- [Derived] Linnemayr S, Huang H, Luoto J, Kambugu A, Thirumurthy H, Haberer JE, Wagner G, Mukasa B. Text Messaging for Improving Antiretroviral Therapy Adherence: No Effects After 1 Year in a Randomized Controlled Trial Among Adolescents and Young Adults. Am J Public Health. 2017 Dec;107(12):1944-1950. doi: 10.2105/AJPH.2017.304089. Epub 2017 Oct 19. PMID 29048966
- [Derived] Patel AR, Lester RT, Marra CA, van der Kop ML, Ritvo P, Engel L, Karanja S, Lynd LD. The validity of the SF-12 and SF-6D instruments in people living with HIV/AIDS in Kenya. Health Qual Life Outcomes. 2017 Jul 17;15(1):143. doi: 10.1186/s12955-017-0708-7. PMID 28716065
- [Derived] Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, Chung MH, Jack W, Habyarimana J, Sadatsafavi M, Najafzadeh M, Marra CA, Estambale B, Ngugi E, Ball TB, Thabane L, Gelmon LJ, Kimani J, Ackers M, Plummer FA. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45. doi: 10.1016/S0140-6736(10)61997-6. Epub 2010 Nov 9. PMID 21071074
- [Derived] Lester RT, Mills EJ, Kariri A, Ritvo P, Chung M, Jack W, Habyarimana J, Karanja S, Barasa S, Nguti R, Estambale B, Ngugi E, Ball TB, Thabane L, Kimani J, Gelmon L, Ackers M, Plummer FA. The HAART cell phone adherence trial (WelTel Kenya1): a randomized controlled trial protocol. Trials. 2009 Sep 22;10:87. doi: 10.1186/1745-6215-10-87. PMID 19772596